CLINICAL TRIAL: NCT04828642
Title: Vitamins C and Vitamin E and Hypertrophy Adaptations to Resistance Traini
Brief Title: Antioxidant Vitaminas and Hypertrophy Adaptations to Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, María Martínez Ferrán, predoctoral researcher, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CIPI/20/209
Record Dates: First submitted 2021-03-11; First posted 2021-04-02 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Hypertrophy
MeSH Terms: conditions — Hypertrophy | interventions — Ascorbic Acid; Vitamin E; Tocopherols

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-control, parallel controlled trial will be conducted.
Who Masked: Participant, Investigator
Masking Description: The provider will produce the supplementation and the placebo with the same aspect, marked with numbers
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplementation group (Active Comparator): Antioxidant vitamins (Vitamin C (1000 mg) + Vitamine E (235 mg))
  Interventions: Dietary Supplement: Vitamin C and vitamin E
- Placebo group (Placebo Comparator): Placebo supplementation with the same aspect as supplementation
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C and vitamin E — 1000 mg 235 mg
  Other Names: Ascorbic acid and tocopherol
  Arms: Supplementation group
Dietary Supplement: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
This investigations aims to investigate whether supplementation with antioxidant vitamins (vitamin C and vitamin E) can influence, enhancing or blocking, the hypertrophic adaptations caused by strength training in sedentary subjects.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-control controlled trial will be conducted. In a previous session volunteers will be interviewed to determine if they meet the inclusion criteria. Will be done two weeks of flushing out other types of supplementation and strenuous physical exercise, along with familiarization with the strength training program and performance tests to be carried out during the rehearsal. Subsequently, it will be a week without exercising to start with the experimental designs. From the start of the trial, participants should avoid physical exercise. strenuous outside the training protocol and if usual, they will only be able to perform one resistance training session per week. Participants should avoid ingesting of foods that contain high amounts of antioxidant compounds: more than two juices of fruits, more than four cups of coffee or tea. Juices with high antioxidant content should be avoided. Alcoholic beverages should also be avoided.

* Group 1 (G1): Antioxidant vitamins (VitC (1000 mg) + VitE (235 mg)) + exercise
* Group 2 (G2): Placebo + exercise A supplementation period of 12 weeks will be carried out. In each period, supplementation with antioxidant vitamins: VitC (1000 mg) + VitE (235 mg) or with placebo.

All participants will ingest the supplementation between 1-3 hours before training, the days of rest in the mornings.

All participants will perform a 12-week strength training protocol. The training session performed in the sharp design will be the first training session in chronic design. Being the baseline (E0) and post-exercise (E1) assessment performed in G1, G2 and G3 also the first evaluation corresponding to the chronic design.

In the middle of the supplementation period (week 6) and at the end, two new evaluations (week 12). Baseline evaluations will be performed prior to an exercise session of week 6 (E2) and at the last exercise session (E3) of the following parameters: performance physique, body composition, micronutrient analysis, muscle ultrasound. I also know conduct post-exercise physical performance assessments Figure 2.

The strength training protocol will be carried out 4 days a week at the facilities sports of the European University. The sessions will be planned by a professional from the Sciences of Physical Activity and Sports. Sessions will be tracked through a diary.

ELIGIBILITY:
Inclusion Criteria:

* Experience in strength training of at least one year

Exclusion Criteria:

* Smokers
* Antioxidant supplementation
* Injuries or diseases

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
DEXA | Week 0
  Evaluation of muscle mass with dual energy X-ray absorptiometry
DEXA | Week 10
  Evaluation of muscle mass with dual energy X-ray absorptiometry
Anthropometry | Week 0
  Evaluation of muscle mass by a ISAK 1 level anthropometrist
Anthropometry | Week 5
  Evaluation of muscle mass by a ISAK 1 level anthropometrist
Anthropometry | Week 10
  Evaluation of muscle mass by a ISAK 1 level anthropometrist
Bioimpedance | Week 0
  Evaluation of muscle mass with an Inbody
Bioimpedance | Week 5
  Evaluation of muscle mass with an Inbody
Bioimpedance | Week10
  Evaluation of muscle mass with an Inbody
DOMS | Week 0
  Delayed onset muscle soreness evaluated with visual analoguic scale (0 no pain- 10 maximal pain)
DOMS | Week 5
  Delayed onset muscle soreness evaluated with visual analoguic scale (0 no pain- 10 maximal pain)
DOMS | Week 10
  Delayed onset muscle soreness evaluated with visual analoguic scale (0 no pain- 10 maximal pain)
Manual dinamometry | Week 0
  Handgrip
Manual dinamometry | Week 5
  Handgrip
Leg dinamometry | Week 0
  Dinamometer
Leg dinamometry | Week 5
  Dinamometer
Leg dinamometry | Week 10
  Dinamometer
RPE | Week 0
  10-point scale (no exertion 0- maximal effort 10)
RPE | Week 5
  10-point scale (no exertion 0- maximal effort 10)
RPE | Week 10
  10-point scale (no exertion 0- maximal effort 10)
1 RM | Week 0
  Bench press and squats
1 RM | Week 5
  Bench press and squats
1 RM | Week 10
  Bench press and squats
Parameters determined by ENCODER | Week 0
  Bench press and squats
Parameters determined by ENCODER | Week 5
  Bench press and squats
Parameters determined by ENCODER | Week 10
  Bench press and squats

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dutra MT, Martins WR, Ribeiro ALA, Bottaro M. The Effects of Strength Training Combined with Vitamin C and E Supplementation on Skeletal Muscle Mass and Strength: A Systematic Review and Meta-Analysis. J Sports Med (Hindawi Publ Corp). 2020 Jan 8;2020:3505209. doi: 10.1155/2020/3505209. eCollection 2020. PMID 31970196
- [Result] Dutra MT, Alex S, Mota MR, Sales NB, Brown LE, Bottaro M. Effect of strength training combined with antioxidant supplementation on muscular performance. Appl Physiol Nutr Metab. 2018 Aug;43(8):775-781. doi: 10.1139/apnm-2017-0866. Epub 2018 Jun 25. PMID 29939770